CLINICAL TRIAL: NCT02006407
Title: A Pilot Study to Evaluate Neurocognitive Injury and Longitudinal Changes in White Matter During Radiation Therapy in Children With Primary Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial closed due to low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCC 2012.117
Record Dates: First submitted 2013-11-26; First posted 2013-12-10 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Brain Tumor, Primary
MeSH Terms: conditions — Brain Neoplasms | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary Brain Tumor (Other): Patients receiving standard cranial radiotherapy will undergo (1) Magnetic Resonance Imaging (MRI) with Diffusion Tensor Imaging (DTI) and (2) Neuro-cognitive testing (CogState-a computerized software testing system that offers various cognitive assessments based on traditional expansive neurocognitive tests) at four timepoints (Baseline, 3 weeks, 6 weeks and 6 months).
  Interventions: Radiation: Cranial Radiotherapy; Device: MRI with Diffusion Tensor Imaging (DTI); Behavioral: Neuro-cognitive Testing (CogState)

INTERVENTIONS:
Radiation: Cranial Radiotherapy — Standard cranial radiotherapy administered dependent upon patient and brain tumor type.
Device: MRI with Diffusion Tensor Imaging (DTI) — Magnetic Resonance Imaging (MRI) with Diffusion Tensor Imaging (DTI)
Behavioral: Neuro-cognitive Testing (CogState) — CogState is a computerized software testing system that offers various cognitive assessments based traditional expansive neurocognitive tests.

SUMMARY:
This is a pilot study to assess the changes in white matter, in the brain, in response to radiation therapy and correlate these changes with later declines in cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (age 6-21) who will receive cranial radiotherapy for brian tumors. This could include but is not limited to: low grade glioma, high grade glioma (to include grade III but not grade IV glioma), germ cell tumors, primitive neuroectodermal tumors, craniopharyngioma, or medulloblastoma.
* Patients should, in the estimate of the treating physician, be anticipated to have a median survival of greater than 1 year.

Exclusion Criteria:

* Patients with previous Central Nervous System (CNS) radiation or or CNS tumors that, in the judgement of the investigators, are likely to undergo progression during or shortly after radiotherapy are excluded.
* Patients with glioblastoma, multiforme, gliosarcoma, diffuse pontine glioma, or other tumors presumed to have expected median survival per the investigators of less than 1 year.
* Patients who require sedation for Magnetic Resonance Imagining (MRI)are excluded.
* Patients at risk for nephrogenic systemic sclerosis will be excluded as a safety precaution due to the contrast used in the scans.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Koschmann, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Brain Tumor
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Brain Tumor
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 14 [8 to 15]
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Change From Baseline in Perpendicular Diffusivity of Water as Measured by Diffusion Tensor Imaging (DTI) at 3 Weeks and at 6 Weeks Post Radiation Therapy.
Description: Descriptive statistics and plots will be used to determine Diffusion Tensor Imaging (DTI) parameters for various regions in the brain. The mean (across subject) change in DTI parameter for a given region, at a given time, will be used to assess white matter injury.
Time Frame: Baseline, 3 weeks, and 6 weeks
Population: Because the outcome measure was CHANGE FROM BASELINE to 3 and 6 weeks, and data were not able to be collected at 3 and 6 weeks, the outcome measure could not be analyzed
Arm/Group | Primary Brain Tumor
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate the Correlation Between Global COGState Scores and the Perpendicular Diffusivity of Water by Diffusion Tensor Imaging at Baseline, 3 Weeks, and 6 Weeks Into Treatment.
Description: Determine the change in cognitive test scores from baseline to time-points early during radiation therapy (3 and 6 weeks) using CogState (a computerized software testing system that offers various cognitive assessments based on expansive neurocognitive tests). Correlate test scores from COGState with changes in Diffusion Tensor Imaging (DTI) at the same timepoints using scatter plots with Pearson and Spearman's correlation coefficients. As a pilot study multiple comparisons will be assessed; however, the working hypothesis is that DTI changes as measured by an increase in diffusivity of water perpendicular to the direction of axonal transport will be measurable even in this acute setting and will correlate with global response as measured on COGState with the sub-domains on executive function anticipated to be most highly correlated.
Time Frame: Baseline, 3 weeks, and 6 weeks
Population: Data can not be accessed due to technical difficulties with the COGState server.
Arm/Group | Primary Brain Tumor
Number analyzed (Participants) | 0

3. Secondary Outcome: Evaluate the Correlation Between Global COGState Scores, Radiation Dose, and the Perpendicular Diffusivity of Water as Measured by Diffusion Tensor Imaging at 6 Months
Description: Determine the change in cognitive test scores from baseline, at 6 months using CogState (a computerized software testing system that offers various cognitive assessments based on expansive neurocognitive tests). Correlate test scores from COGState with changes in Diffusion Tensor Imaging (DTI) at the same timepoints (Baseline and 6 months) using scatter plots with Pearson and Spearman's correlation coefficients. As a pilot study multiple comparisons will be assessed; however, the working hypothesis based upon results in adults treated with radiation therapy is that DTI changes as measured by an increase in diffusivity of water perpendicular to the direction of axonal transport will correlate with changes in global response as measured on COGState with the sub-domains on executive function most highly correlated. In addition, these regional changes in DTI will be directly related to the radiation doses received in these regions.
Time Frame: 6 months
Population: Data can not be accessed due to technical difficulties with the COGState server.
Arm/Group | Primary Brain Tumor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected from the time of the initial study intervention through the 12 month post baseline visit.
Description: Only events related to the study intervention (MRI and Neuro-cognitive Testing) were reported. No adverse events related to these interventions were reported.
Arm/Group | Primary Brain Tumor
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes